CLINICAL TRIAL: NCT05331209
Title: Acupuncture With or Without Self-acupressure for Hot Flashes in Post-oophorectomy Patients With BRCA Mutations: A Prospective, Randomized Controlled Trial
Brief Title: Acupuncture With/Without Self-acupressure for Post-oophorectomy Hot Flashes in BRCA Carriers
Acronym: BRCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Noah Samuels, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRCA-ACP.2022
Record Dates: First submitted 2022-04-09; First posted 2022-04-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Hot Flashes; Menopause Surgical
Keywords: acupuncture; acupressure; hot flashes; surgical menopause; quality of life
MeSH Terms: conditions — Hot Flashes | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, open, randomized, add-on
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture only (Active Comparator): Acupuncture treatments will take place at a frequency of once per week, with each session lasting between 30 to 45 minutes. At each session patients will be re-assessed by the study acupuncturist, with acupuncture points individualized in accordance with the principles of traditional Chinese medicine. At the same time, acupuncturists will include a set group of acupuncture points which have been used in the research of hot flashes: HT-6, Kid-3, Liv-3, SP-6.
  Interventions: Other: Acupuncture; Other: Acupuncture-Acupressure
- Acupuncture-Acupressure (Active Comparator): Patients randomly allocated to the acupuncture-acupressure arm of the study will first be treated by the study acupuncturist in accordance with the protocol described in the Acupuncture arm of the study. At the end of the first session, patients in this group will be taught by the study acupuncturist to self-treat at home with acupressure, on the acupressure points PC-7, ST-36, SP-9. Self-acupressure sessions will last between 3-5 minutes each, and will take place 3-4 times each day. At subsequent acupuncture treatments patients will receive reinforcement and guidance to ensure the fidelity of the self-acupuncture treatments
  Interventions: Other: Acupuncture; Other: Acupuncture-Acupressure

INTERVENTIONS:
Other: Acupuncture — Weekly acupuncture treatments, for 8 weeks (8 treatments)
Other: Acupuncture-Acupressure — Weekly acupuncture, for 8 weeks, with daily self-acupressure by the patient at home.

SUMMARY:
Risk-reducing surgery with salpingo-oophorectomy (RRSO) is the standard recommended treatment for all female carriers of BRCA genes 1 and 2. The post-surgical menopause induced is invariably accompanied by hot flashes and other symptoms, which can severely impair quality of life and function. Hormone-replacement therapy (HRT) is the standard conventional treatment for these symptoms, though these drugs do not always provide adequate relief and many patients either cannot receive them due to a diagnosis of breast cancer or hypercoagulable state; or are unwilling to take them due to their concern about the associated increased risk for developing hormone-induced breast cancer.

Acupuncture and acupressure have been researched extensively and shown to be both safe and effective in reducing hot flashes in post-menopausal patients and in those with breast cancer receiving anti-hormonal drugs.

The present study will examine the effectiveness of acupuncture, with/without self-acupressure, on 200 post- RRSO patients who suffer from at least 5 hot flashes per day, including those treated with HRT. All participants will receive 8 weekly treatments with acupuncture, and then randomly assigned to receive (or not) self-administered acupressure, to be performed daily at home. The response to the study interventions will be assessed using daily Hot Flash Scores, the Menopause Specific Quality of Life (MenQoL) and Measure Yourself Concerns and Wellbeing (MYCAW) questionnaires (at baseline; at the end of the 8-week intervention; and at 16 weeks). The safety of the study treatments will be assessed throughout.

ELIGIBILITY:
Inclusion Criteria:

* Female carriers of the BRCA 1 and 2 genes
* age ≥ 25 years
* after risk-reducing salpingo-oophorectomy
* reporting ≥ 5 hot flashes per day

Exclusion Criteria:

* Patients not fulfilling the study inclusion criteria will be excluded from participation

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study interventions will be provided to female patients who are carriers of the BRCA 1 and 2 genes who suffer from hot flashes following risk-reducing salpingo-oophorectomy (RRSO). The intervention is not relevant for patients of other genders.
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hot Flash Score - baseline to 8 weeks | From baseline (at study recruitment) to end of intervention (8 weeks)
  Hot Flash Score will be calculated by the following equation: Mean number daily hot flashes X mean severity of symptoms (Hot flash severity: 1 - mild; 2 - moderate; 3 - severe)

SECONDARY OUTCOMES:
Hot Flash Score - 8 to 16 weeks | From end of study intervention (at 8 weeks) to end of post-intervention period (16 weeks)
  Hot Flash Score will be calculated by the following equation: Mean number daily hot flashes X mean severity of symptoms (Hot flash severity: 1 - mild; 2 - moderate; 3 - severe)
Menopause Specific Quality of Life Questionnaire (MenQOL) | Baseline; End of intervention (8 weeks); Post-treatment follow-up (16 weeks)
  The MenQoL study tool assesses health-related quality of life in the immediate postmenopausal period. The tool contains 29 items from four menopausal symptom domains, as experienced over the last month: vasomotor, psychosocial, physical, and sexual. Means are computed for each subscale by dividing the sum of the items in the domain by the number of items within that domain; the final score ranges from 1 to 8.41 For the present study, the questionnaire was translated from English into Hebrew by 2 fully bilingual medical professionals, and then back-translated by 2 other fully bilingual medical professionals, in accordance with acceptable measurement translation methods.
Measure Yourself Concerns and Wellbeing (MYCAW) | Baseline; End of intervention (8 weeks); Post-treatment follow-up (16 weeks)
  The MYCAW (Appendix 2) asks respondents at baseline to list their two main concerns, scoring their severity from a range of 0 (of no concern) to 6 (of greatest concern). Patients are then asked to score the quality of their present level of well-being, from a score of 0 ("as good as it could be") to 6 ("as bad as it could be"). At the follow-up completion of the tool patients are asked once again to score the two primary concerns (listed at baseline), as well as their current perceived level of wellbeing. The follow-up questionnaire then asks respondents to answer two open-ended questions: the first about "other issues related to your health"; and the second, "what has been the most important aspect (of the treatment program) for you?".

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Integrative Complementary Medicine, Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No